CLINICAL TRIAL: NCT05044351
Title: Autofluorescence-guided Hemithyroidectomy in a Low-volume, Non-parathyroid Insitution: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Responsible Party: Principal Investigator, Ali Abood, MD, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Autofluorescence2.0
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Autofluorescence; Thyroidectomy; Autotransplantation

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider
Masking Description: Patients and related health care staff will be blinded for the allocated intervention until the day of surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (A): NIRAF-assisted surgery (Experimental): Patients undergoing NIRAF-assisted hemithyroidectomy
  Interventions: Device: Fluobeam LX
- (B): Conventional surgery (Active Comparator): Patients undergoing conventional hemithyroidectomy without NIRAF-assistance
  Interventions: Other: Conventional surgery without NIRAF assistance

INTERVENTIONS:
Device: Fluobeam LX — See arm description
  Arms: (A): NIRAF-assisted surgery
Other: Conventional surgery without NIRAF assistance — Patients undergoing conventional hemithyroidectomy without NIRAF-assistance
  Arms: (B): Conventional surgery

SUMMARY:
Parathyroid damage and inadvertent excision unfortunately happens frequently in thyroid surgery. The use of near-infrared autofluorescence (NIRAF) intraoperatively, seems to be helpful in terms of parathyroid identification and preservation.

In order to cover every aspect of the impact of NIRAF in thyroid surgery, an evaluation in low-volume, non-parathyroid centers is needed:

Aim: To investigate the impact of NIRAF on hemithyroidectomy by evaluating parathyroid identification, damage and the rate of inadvertent parathyroid excision in a low-volume, non-parathyroid institution.

DETAILED DESCRIPTION:
Patients referred for hemithyroidectomy will be randomized to either:

(A) NIRAF-assisted hemithyroidectomy (Fluobeam LX) or (B) Conventional hemithyroidectomy. PTH and ionized calcium will assessed preoperatively, on postoperative day 1 (POD1) and one month following surgery. Parathyroid identification rates, rates of autoimplantation and inadvertently excised parathyroid glands will be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for thyroid lobectomy
* Age > 18
* Able to understand patient information
* Able to give informed consent

Exclusion Criteria:

* Completion lobectomy
* Need for accelerated surgery
* Age < 18
* Unable to understand patient information
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Parathyroid gland identification rate | Will be assessed at the time of surgery

SECONDARY OUTCOMES:
Rate of inadvertent parathyroid excision | Will be assessed one month following surgery
Rate of autotransplantation | Will be assessed at the time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Regional Hospital West Jutland, Holstebro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abood A, Rolighed L, Ovesen T, Madsen SH, Vestergaard P, Triponez F. Autofluorescence-guided hemithyroidectomy in a low-volume thyroid institution with no experience in parathyroid surgery: randomized clinical trial. Br J Surg. 2024 Apr 3;111(4):znae075. doi: 10.1093/bjs/znae075. PMID 38573333